CLINICAL TRIAL: NCT04302519
Title: Clinical Study of Novel Coronavirus Induced Severe Pneumonia Treated by Dental Pulp Mesenchymal Stem Cells
Brief Title: Novel Coronavirus Induced Severe Pneumonia Treated by Dental Pulp Mesenchymal Stem Cells
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CAR-T (Shanghai) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KT005HB001
Record Dates: First submitted 2020-02-27; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Dental pulp mesenchymal stem cells were injected intravenously
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulp mesenchymal stem cells (Experimental): 1. 3, 7 days to increase the injection of mesenchymal stem cells
  Interventions: Biological: Dental pulp mesenchymal stem cells

INTERVENTIONS:
Biological: Dental pulp mesenchymal stem cells — On the basis of clinical standard treatment, the injection of dental mesenchymal stem cells was increased on day 1, 3 and 7 of the trial.

SUMMARY:
Evaluation of novel coronavirus induced severe pneumonia by dental pulp mesenchymal stem cells

DETAILED DESCRIPTION:
Open, single center, single arm test design. Plan to enroll 24 subjects. On the basis of clinical standard treatment, the injection of dental mesenchymal stem cells was increased on day 1, 3 and 7 of the trial.

Injection dose: 1.0x106 cells /kg. Injection method: slowly and quietly drop 50 mL of normal saline, then the endodontic mesenchymal stem cell injection (after 60 min), and then 50 mL of normal saline.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18, age ≤ 75, gender unlimited;
* 2. novel coronavirus diagnosed severe pneumonia and confirmed no effective treatment plan. (severe patients meet any of the following: (1) respiratory distress, RR > 30 times / minute; (2) resting state, oxygen saturation is less than 93%; (3) arterial oxygen partial pressure (PaO2) / oxygen inhalation (FiO2) is less than 300 mmHg (1mm Hg=0.133 kPa).
* 3. Those who voluntarily participate in the clinical study and can cooperate with researchers to carry out the study, and the patients themselves or their legal representatives voluntarily sign the informed consent.

Exclusion Criteria:

* 1. Patients with autoimmune diseases in the past or screening;
* 2. Those who have serious basic diseases that affect their survival, including: malignant tumor, hematopathy, malignant fluid, active hemorrhage, severe malnutrition, etc. which have not been controlled and can not be removed due to multiple metastasis;
* 3. Known or self-reported HIV or syphilis infected persons;
* 4. Have participated in stem cell clinical research;
* 5. Pregnant or lactating women or those who have fertility plans in the past year;
* 6. The estimated life cycle is less than 48 hours;
* 7. Those who participated in other clinical trials within 3 months before screening;
* 8. Other conditions that the researcher thinks are not suitable for participating in the experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-03-05 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Disppear time of ground-glass shadow in the lungs | 14 days
  Kaplan-meier method was used to calculate the median glassy shadow time in all subjects

SECONDARY OUTCOMES:
Absorption of Lung shadow absorption by CT Scan-Chest | 7, 14, 28 and 360 days
  Kaplan-meier method was used to calculate the median lung shadow absorption of all subjects on 7, 14, 28, and 360 days
Changes of blood oxygen | 3, 7 and 14 days
  T test was used to compare the blood oxygen values of each subject at day 3, 7 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Liwei cheng, doctor, Study Director — Research office of wuhan renmin university

IPD SHARING:
Plan to Share IPD: No